CLINICAL TRIAL: NCT07247227
Title: Sugemalimab Plus Platinum-based Chemotherapy as First-line Therapy for Patients With Locally Advanced and Metastatic Non-small Cell Lung Cancer (NSCLC) in a Real-world Setting: a Single-arm, Multi-center Study
Brief Title: Real-world First-line Sugemalimab-Chemotherapy in Advanced NSCLC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking Union Medical College (Other)
Responsible Party: Principal Investigator, Junling Li, professor, Peking Union Medical College
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCC3980
Record Dates: First submitted 2025-11-17; First posted 2025-11-25 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: NSCLC
Keywords: sugemalimab; NSCLC
MeSH Terms: interventions — sugemalimab; Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- stage IV NSCLC. (Experimental): Sugemalimab 1200mg plus 4-6 cycles of platinum-based chemotherapy
  Interventions: Drug: Sugemalimab and Chemotherapy
- stage III NSCLC. (Experimental): sugemalimab+platinum-based chemotherapy in stage III NSCLC.
  Interventions: Drug: Sugemalimab and Chemotherapy

INTERVENTIONS:
Drug: Sugemalimab and Chemotherapy — Sugemalimab 1200mg plus 4-6 cycles of platinum-based chemotherapy as first-line therapy, followed by Sugemalimab 1200mg to 35 cycles, or until disease progression, or ICF withdrawn by participants, or death or unacceptable toxicity.

SUMMARY:
This single-arm, multi-center study is to evaluate Sugemalimab plus platinum-based chemotherapy as first-line therapy for patients with locally advanced and metastatic NSCLC in a real-world setting.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years.
2. Patients voluntarily join the study and sign an informed consent form for the study.
3. ECOG PS score 0-3 (patients with PS score 2-3 would be enrolled if due to the tumor disease and anticipated to be improved at investigators' decision).
4. Histologically documented, stage III, IV non-Small Cell Lung Cancer (according to version 8th of the International Association for the Study of Lung Cancer Staging Manual in Thoracic Oncology) and previously untreated systematically(excluding local therapy for local lesions or symptomatic relief, palliative radiotherapy, intervention, intrathecal injection, nerve block, etc.).
5. Patients with stage III NSCLC who are not suitable for surgery at a multidisciplinary discussion or investigators' assessment.
6. Patients with at least one measurable target lesion by CT scan/MRI (RECISTv1.1).
7. Patients with active brain metastases and liver metastases could be enrolled (Concurrent radiotherapy, intervention, dehydration, and other local treatment are permitted).
8. Interstitial pneumonia, drug-induced pneumonia, radiation pneumonitis requiring steroid therapy, or active pneumonia with clinical symptoms of grade 2, can be included after symptomatic treatment until recovery to grade 0-1.
9. Fertile men and women of childbearing age must agree to take effective contraceptive measures from signing the main informed consent until 180 days after the last dose of the study drug. Women of childbearing potential include premenopausal women and women within 2 years of menopause. Females of childbearing potential must have a negative pregnancy test ≤ 7 days prior to the first dose of study drug.

Exclusion Criteria:

1. All patients carry activating mutations of EGFR, ALK, ROS1, and RET. (No more mutation test needed).
2. Small cell lung cancer (including patients with mixed small cell lung cancer and non-small cell lung cancer).
3. Histopathologically or cytopathologically confirmed non-NSCLC.
4. Any prior treatment of antibody/drug that targets T-cell coregulatory proteins (not limited to CTLA-4 inhibitors or other agents targeting T cells).
5. Any tumor history within the past 5 years prior to the start of treatment in this study (except cured cervical carcinoma in situ, cured basal cell carcinoma, and bladder epithelial tumors with surgical resection alone and at least 5 consecutive years of disease-free survival).
6. Patients with active, unstable systemic disease, active infection, uncontrolled hypertension, heart failure (NYHA class >= II), unstable angina pectoris, acute coronary syndrome, severe arrhythmia, severe liver, kidney, or metabolic diseases, HIV infection.
7. Pregnant or lactating women.
8. Systemic anti-tumor therapy planned within 4 weeks before first-line treatment or during medication after enrollment, including cytotoxic therapy, signal transduction inhibitors, immunotherapy (with the exception of thymosin, lentinan, and other immunomodulator therapy).
9. Major surgical treatment, incisional biopsy, or significant traumatic injury within 28 days before 1st line therapy.
10. Participation in other anti-tumor drug clinical trials within 4 weeks before first-line therapy.
11. Active, known, or suspected autoimmune diseases. Vitiligo and Type I diabetes mellitus with no systemic treatment are allowed. Residual hypothyroidism caused by autoimmune thyroiditis requiring only hormone replacement therapy is allowed.
12. With known mental illness, alcoholism, drug abuse, or other factors which may cause termination of this study, affect the safety of subjects, or collection of data and samples.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2023-10-10 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
rw-PFS | From enrollment to the end of treatment at 1 year
  rw-PFS, defined as the time from the start of 1st line treatment to tumor progression or death, which occurs first

SECONDARY OUTCOMES:
TTF | From enrollment to the end of treatment at 1 year
  time from the start of the first dose of first-line therapy to treatment failure due to any cause.
OS | From enrollment to the end of treatment at 1 year
  OS defined as the time from the start of treatment to death from any cause.
Objective response rate (ORR) | From enrollment to the end of treatment at 1 year
  the proportion of patients with a complete response (CR) or a partial response (PR), as assessed by RECIST version 1.1 Subjects with measurable disease and CR or PR determined at least 4 weeks after initial CR or PR would be considered responders.
DCR | From enrollment to the end of treatment at 1 year
  the proportion of patients with disease control (CR,PR or SD), as assessed by RECIST version 1.1
DOR | From enrollment to the end of treatment at 1 year
  For subjects who demonstrated CR or PR, duration of response (DOR) is defined as the time from first documented evidence of CR or PR until disease progression or death
Safety, number of participants with treatment-related adverse events (AEs) | From enrollment to the end of treatment at 1 year
  Including treatment-emergent adverse reactions (AEs), drug-related AEs, serious adverse reactions (SAEs), and drug-related SAEs
12-month, 18-month, and 24-month overall survival (OS) rates | Up to 24 months from treatment initiation (with OS rates assessed at 12, 18, and 24 months)
  The 12-, 18-, and 24-month overall survival (OS) rates are defined as the proportions of patients who are alive at 12, 18, and 24 months after treatment initiation, respectively.

CONTACTS AND LOCATIONS:
Locations (1):
- cancer hospital， Chinese Academy of medical sciences and Peking union medical college, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No